CLINICAL TRIAL: NCT01811173
Title: The Clalit Comprehensive-Care for Multimorbid Adults Project
Brief Title: Comprehensive-Care for Multimorbid Adults Effectiveness Study
Acronym: CCMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCMAP
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Disease
Keywords: multimorbidity; primary care; physician - nurse team; proactive monitoring; support for self-care; primary caregiver
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nurse-physician comprehensive care (Experimental): Comprehensive self management support and care coordination by a nurse-primary care physician team
  Interventions: Other: Nurse-physician comprehensive care
- Usual care survey control group (No Intervention): Patients will receive usual primary care and asked to complete questionnaires on four time points throughout the study
- Usual care blinded control group (No Intervention): Patients will receive usual primary care.

INTERVENTIONS:
Other: Nurse-physician comprehensive care — Components of the intervention include:
  1. Complete assessment of the patient's and family's needs conducted by the nurse.
  2. Comprehensive treatment program developed by the nurse and in consultation with the primary care physician.
  3. "Multimorbid care plan" integrating all care aspects.
  4. "Action Plan" for patients, supporting self management
  5. Proactive monitoring according to the plan.
  Arms: Nurse-physician comprehensive care

SUMMARY:
This study is intended to examine whether directed care of a nurse working jointly with the patient's primary care physician, including a comprehensive assessment, creation of a tailored care plan, proactive follow-up, self management support and caregiver support and care coordination, can reduce hospital admissions for patients with multiple chronic conditions.

DETAILED DESCRIPTION:
Patients with multi-morbidities pose a significant challenge for healthcare organizations because they require continuity of care among a wide range of long-term therapeutic paradigms for many different types of diseases. The current study is based on a treatment model entailing a nurse-primary care physician team to provide care for patients with multiple morbidities.

Patients in the intervention group who agreed and signed the consent form to participate in the study will receive treatment by the physician - nurse team in accordance with the components of the Clalit's Comprehensive Care for Mutlimorbid Adults Project model. Components of the intervention include:

1. Comprehensive assessment of the patient's and family's needs
2. Coordinated care plan based on integrated care guides
3. "Multimorbid Action Plan" for patients
4. All-inclussive patient centered care and caregiver support
5. Proactive monitoring according to the plan.

Patients in the control groups will receive usual care in their primary care clinics. The Usual Care Survey control group will complete study questionnaires at 6, 12 and 24 months after enrollement.

The Usual Care Blinded group will be assessed only retrospectively based on deidentified information from Clalit's admistrative databases.

ELIGIBILITY:
Inclusion Criteria:

* ACG system high risk probabilty score - 4% Highest Risk Score
* Age 18 and older
* 2 or more chronic conditions

Exclusion Criteria:

* Patients already included in a controlled disease management program (e.g., COPD disease management and telehealth).
* Participation in any medical research.
* Confined to bed.
* Inpatient nursing care, nursing homes.
* Kidney, liver or heart transplant patients.
* Active (receipt of oncology chemotherapy , radiotherapy or other oncology treatment during the past 3 years).
* Dialysis patients.
* Clalit Healthcare Services employees.
* Patients with major active mental illness, such as schizophrenia.
* Cognitive failure.
* Non Hebrew speaking patients without Hebrew speaking primary informal caregiver.
* Bedridden patients
* Housebound patients

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Percent change in admissions for ambulatory care sensetive conditions | At enrollment and within 12 months and 24 months after enrollment
  Ambulatory Care Sensitive Conditions will be defined by ICD-9 codes, based on the classification published by: Ansari, Barbetti, Carson, Auckland, & Cicuttini, 2003 (adapted from Weissman JS, Gatsonis C, Epstein AM ,1992; Millman M, ed. 1993)

SECONDARY OUTCOMES:
Emergency 30-day readmissions | 30 days post an index admission
  Emergency readmissions are defined as an urgent (via the Emergency Room) admission of one night or longer, following an index admission that lasted 2 nights or longer, in the prior 30 days.

OTHER OUTCOMES:
Change in SF-12 Physical and Menal component scores | At enrollment and 6, 12, and 24 months after enrollment
  Change in Physical and Menal Component scores of the SF-12 measure, as completed by patients through patient interviews

CONTACTS AND LOCATIONS:
Overall Officials: Ran D Balicer, PhD, Principal Investigator — Clalit Research Institute, Clalit Health Services
Locations (13):
- Israel (13):
  - Ashdod A, Ashdod
  - Ashdod D, Ashdod
  - Azur, Azor
  - Arlozorov, Bat Yam
  - Hashikma, Bat Yam
  - Ramat Yosef, Bat Yam
  - Sokolov, Bat Yam
  - Halutz, Hulon
  - Shikun Ammi, Hulon
  - Lod Center, Lod
  - Ramla Ztafon, Ramla
  - Balfur, Rishon LeZiyyon
  - Migdal HaIr, Rishon LeZiyyon

REFERENCES:
- [Derived] Cohen-Stavi CJ, Giveon S, Key C, Molcho T, Balicer R, Shadmi E. Guideline deviation and its association with specific chronic diseases among patients with multimorbidity: a cross-sectional cohort study in a care management setting. BMJ Open. 2021 Jan 11;11(1):e040961. doi: 10.1136/bmjopen-2020-040961. PMID 33431488
- [Derived] Steinman MA, Low M, Balicer RD, Shadmi E. Impact of a nurse-based intervention on medication outcomes in vulnerable older adults. BMC Geriatr. 2018 Sep 6;18(1):207. doi: 10.1186/s12877-018-0905-1. PMID 30189846